CLINICAL TRIAL: NCT01056848
Title: International, Multicenter Study of a Twenty-eight Week, Open-label, Titrated Oral Lixivaptan Administration in Patients With Chronic Hyponatremia: Extension to Studies CK-LX3401, 3405, and 3430
Status: Completed | Type: Observational
Sponsor: CardioKine Inc. (Industry)
Collaborators: Cardiokine Biopharma, LLC (Industry); Biogen (Industry)
Responsible Party: Cesare Orlandi, MD, Cardiokine Biopharma, LLC
Other Study IDs: CK-LX3431
Record Dates: First submitted 2010-01-22; First posted 2010-01-26 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Hyponatremia With Normal Extracellular Fluid Volume; Hyponatremia With Excess Extracellular Fluid Volume
Keywords: Euvolemic Hyponatremia; Hypervolemic Hyponatremia; SIADH; Serum Sodium
MeSH Terms: conditions — Inappropriate ADH Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- CK-LX3401: Patients with euvolemic or hypervolemic hyponatremia and who were enrolled in a randomized, blinded, placebo-controlled Phase III lixivaptan study of hyponatremia.
- CK-LX3405: Patients with euvolemic or hypervolemic hyponatremia and who were enrolled in a randomized, blinded, placebo-controlled Phase III lixivaptan study of hyponatremia
- CK-LX3430: Patients with euvolemic or hypervolemic hyponatremia and who were enrolled in a randomized, blinded, placebo-controlled Phase III lixivaptan study of hyponatremia

SUMMARY:
To evaluate the overall safety and continued efficacy of oral lixivaptan capsules in subjects with euvolemic and hypervolemic hyponatremia

DETAILED DESCRIPTION:
Phase I and Phase II clinical trials have demonstrated that lixivaptan may play an important role in treating hyponatremia and the signs and symptoms of water retention associated with HF, LCWA and SIADH. Lixivaptan was previously evaluated in disease states characterized by hyponatremia with euvolemia (SIADH) and hyponatremia combined with fluid overload (HF, LCWA). Lixivaptan demonstrated correction in serum sodium concentration together with marked aquaresis in patients with hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women 18 years of age or older
2. Ability to provide informed consent or assent
3. Prior participation in a lixivaptan hyponatremia trial with evidence of continued need or desire for therapy

Exclusion Criteria:

1. A current medical condition where long-term treatment with an aquaretic agent may present an undue risk to the patient
2. Hyponatremia which is acute, reversible, artificial or due to conditions not associated with vasopressin excess or likely to respond to aquaretic therapy
3. Hyponatremia due to reversible medical condition or therapy
4. Conditions associated with an independent imminent risk of morbidity and mortality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with euvolemic or hypervolemic hyponatremia and who were enrolled in a randomized, blinded, placebo-controlled Phase III lixivaptan study of hyponatremia (CK-LX3401, CK-LX3405, or CK-LX3430)
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2010-01; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
To assess the safety of long-term lixivaptan use in patients who were previously enrolled in one of the 3 Phase III trials. | 28 weeks

SECONDARY OUTCOMES:
To demonstrate that after open-label lixivaptan treatment: improvements in the time to complete the TMT-B will be maintained compared to baseline, and improvements in the Medical Outcomes Survey will be maintained compared to baseline. | 28 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Torrance Clinical Research, Lomita, California
  - Innovative Research of West Florida, Clearewater, Florida
  - Fleming Island Center for Clinical Research, Fleming Island, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Millenium Psychiatric Associates, LLC, Creve Cour, Missouri
  - Internal Medical Associates of Grand Island, PC, Grand Island, Nebraska